CLINICAL TRIAL: NCT07123389
Title: Impact of Family Functioning and Peer Pressure on Nicotine Dependence: A Cross-sectional Study Among Medical Students in South Punjab, Pakistan
Brief Title: Family and Peer Influences on Nicotine Dependence in Medical Students of South Punjab
Status: Completed | Type: Observational
Sponsor: Nishtar Medical University (Other)
Responsible Party: Principal Investigator, Fakiha Sultana Malik, Medical Student, Nishtar Medical University
Other Study IDs: 8975/NMU
Record Dates: First submitted 2025-07-24; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Nicotine Dependence; Tobacco Use Disorder; Family Functioning; Peer Influence
Keywords: Tobacco Use Disorder; Smoking; Medical Students; Family Relations; Peer Influence; Nicotine
MeSH Terms: conditions — Tobacco Use Disorder; Smoking

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Medical Students in South Punjab: Students enrolled at medical colleges in South Punjab, Pakistan who consent to participate. They will complete a structured, self-administered questionnaire assessing nicotine dependence (FTND), family functioning (FAD-GF), and peer pressure, along with basic demographic information.

SUMMARY:
The goal of this cross-sectional observational study is to assess the impact of family functioning and peer pressure on nicotine dependence in medical students enrolled at medical colleges in South Punjab, Pakistan (both male and female; aged 18 and older). The main questions it aims to answer are:

Does family dysfunction contribute to higher nicotine dependence in medical students? Does peer pressure intensify the effect of family dysfunction on nicotine dependence? Are there gender or academic year differences in smoking status and peer pressure?

If there is a comparison group:

Researchers will compare students from functional families vs. dysfunctional families to see if nicotine dependence differs, especially under the influence of peer pressure.

Participants will:

Complete a structured, self-administered questionnaire which includes:

The Fagerstrom Test for Nicotine Dependence (FTND) to assess nicotine addiction severity.

The Family Assessment Device-General Functioning (FAD-GF) to evaluate family functioning.

The Peer Pressure Scale to identify direct and indirect peer pressure. Provide demographic information (age, gender, year of study, smoking status) for descriptive and comparative analyses.

ELIGIBILITY:
Inclusion Criteria:

* Medical students currently enrolled in public or private medical colleges in South Punjab, Pakistan
* Aged 18 years or older
* Voluntarily consent to participate in the study

Exclusion Criteria:

* Refusal to provide informed consent
* Absence or unavailability at the time of data collection
* Incomplete questionnaire or failure to complete the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will recruit medical students enrolled at public and private medical colleges across South Punjab, Pakistan. Participants will be young adults aged 18 and above who are pursuing their Bachelor of Medicine, Bachelor of Surgery (MBBS) degrees. The population will consist of students from all academic years and diverse socioeconomic backgrounds. Medical students were selected due to their future role as healthcare providers and their unique stressors, making them an important group for understanding the interplay of family functioning, peer pressure, and nicotine dependence.
Sampling Method: Non-Probability Sample
Enrollment: 366 (Actual)
Dates: Start 2025-05-13 (Actual); Primary Completion 2025-07-02 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Nicotine Dependence Score as assessed by the Fagerström Test for Nicotine Dependence (FTND) | Day 1
  Primary Outcome: Nicotine Dependence
  The primary outcome of this study is the level of nicotine dependence among medical students, measured using the Fagerström Test for Nicotine Dependence (FTND). The FTND provides a continuous score ranging from 0 to 10, based on six items. Three of these items are yes/no questions, scored as 0 (No) and 1 (Yes). The remaining three are multiple-choice questions, scored from 0 to 3. The scores from all six items are summed to calculate the total dependence score.
  Classification of Nicotine Dependence:
  0-2: Very Low
  3-4: Low
  5: Moderate
  6-7: High
  8-10: Very High
  This continuous FTND score will be used to assess the impact of family functioning and peer pressure on the severity of nicotine addiction.

SECONDARY OUTCOMES:
Prevalence of Dysfunctional Family Functioning as assessed by the Family Assessment Device-General Functioning (FAD-GF) | Day 1
  To evaluate the relationship between family functioning and nicotine dependence, the proportion of medical students reporting dysfunctional family functioning will be assessed. Participants will be provided with the Family Assessment Device - General Functioning subscale (FAD-GF), which includes 12 items designed to measure overall family functioning. Each item will be rated on a 4-point Likert scale, ranging from 1 (Strongly Agree) to 4 (Strongly Disagree). Negatively worded items will require reverse coding to ensure scoring consistency, as higher scores will indicate poorer family functioning.
  A cutoff mean score of 2.00 will be used to classify family functioning:
  Mean score ≥ 2.00: Indicative of dysfunctional or unhealthy family functioning
  Mean score < 2.00: Indicative of functional or healthy family functioning
  This classification will allow examination of the association between family functioning status and the severity of nicotine dependence, as measured by
Prevalence of Peer Pressure Exposure as assessed by the Peer Pressure Scale | Day 1
  Peer pressure will be assessed using the Indicators of Peer Pressure adopted from Subramaniam et al. The questionnaire will contain six questions divided into direct and indirect peer pressure. Students will be asked to answer 'yes' or 'no' to each question. There will be three questions assessing direct peer pressure and three assessing indirect peer pressure. Students who answer 'yes' to any question will be considered to have experienced peer pressure, while those who respond 'no' to all questions will be classified as free from peer pressure.

CONTACTS AND LOCATIONS:
Locations (1):
- Nishtar Medical University, Multan Khurd, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-30): https://cdn.clinicaltrials.gov/large-docs/89/NCT07123389/Prot_SAP_000.pdf